CLINICAL TRIAL: NCT06299982
Title: A Multicenter,Randomized,Phase 3 Trial to Evaluate the Efficacy and Safety of Recombinant Anti-IL-17A Humanized Monoclonal Antibody in Chinese Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: An Phase III Study of Recombinant Anti-IL-17A Humanized Monoclonal Antibody in Chinese Participants With PsO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-608-PsO-III-02
Record Dates: First submitted 2024-02-28; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: Plaque Psoriasis Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 608 160 mg W0+80 mg Q2W (Experimental): Participants will receive starting dose of 160 milligrams (mg) 608 at week 0 followed by 80mg 608 once every two weeks (Q2W) by subcutaneous injection for 12 weeks.
  Interventions: Drug: 608 Q2W
- 608 160 mg Q4W (Experimental): Participants will receive 160 milligrams 608 once every four weeks (Q4W) by subcutaneous injection for 12 weeks.
  Interventions: Drug: 608 Q4W

INTERVENTIONS:
Drug: 608 Q2W — 608 160 mg at week 0 + 80 mg Q2W (5 cycles)
  Arms: 608 160 mg W0+80 mg Q2W
Drug: 608 Q4W — 608 160 mg Q4W (3 cycles)
  Arms: 608 160 mg Q4W

SUMMARY:
The purpose of this study is to examin the efficacy and safety of the study drug recombinant anti-IL-17A humanized monoclonal antibody in Chinese participants with moderate-to-severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, both male and female.
* Diagnosis of plaque psoriasis according to the Chinese Guideline for the Diagnosis and Treatment of Psoriasis (2018).

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and/or guttate psoriasis) .
* Other inflammatory diseases.
* Active autoimmune diseases.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a ≥75% Improvement in Psoriasis Area and Severity Index (PASI 75) | At Week 12
Percentage of Participants With a Static Physician Global Assessment (sPGA) Score of Clear (0) or Minimal (1) With at Least a 2 Point Improvement | At Week 12

SECONDARY OUTCOMES:
Percentage of Participants Achieving a ≥90% Improvement in Psoriasis Area and Severity Index (PASI 90) | At Week 12
Percentage of Participants Achieving a ≥100% Improvement in Psoriasis Area and Severity Index (PASI 100) | At Week 12
Percentage of Participants Achieving a Static Physician Global Assessment (sPGA) Score of Clear (0) | At Week 12
Adverse events (AE) | 20 weeks